CLINICAL TRIAL: NCT03677219
Title: An Educational Video to Address Parental Concern in Lumbar Puncture Consent: A Randomized Control Trial
Brief Title: Lumbar Puncture Video Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ash Singhal, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H14-00981
Record Dates: First submitted 2018-01-17; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Consent
Keywords: consent; lumbar puncture; pediatric; video

STUDY DESIGN:
Intervention Model Description: Parents are randomized to either view an educational video or not
Who Masked: Participant, Care Provider
Masking Description: The caregiver obtaining consent for lumbar puncture does not know if the parent will be randomized to see the video; the parent is not aware they may be randomized to see a video when they respond to the first survey about their concerns.

ARMS (2):
- Control (No Intervention): Parents in this arm receive the standard lumbar puncture consent discussion and answer a survey about their concerns, and do not view an educational video.
- Video (Experimental): Parents in this arm receive the standard lumbar puncture consent discussion and answer a survey about their concerns, then view a 2 minute educational video and respond to a second survey.
  Interventions: Other: Educational Video

INTERVENTIONS:
Other: Educational Video — The educational video is a 2 minute video depicting a live lumbar puncture on an infant interwoven with animations of the relevant anatomy.
  Arms: Video

SUMMARY:
The purpose of this study is to improve the lumbar puncture (LP) consent process for pediatric patients. Though a commonly performed and safe procedure, LP can be anxiety-provoking for parents. By using an educational video on a handheld device at the time of consent, we hope to improve parent understanding and comfort with the procedure.

DETAILED DESCRIPTION:
Introduction: Lumbar puncture is a safe procedure commonly performed on pediatric patients for a variety of indications. Parents are informed of and consented to this procedure, but are often left with concerns and doubts. There are no published studies of the nature of the concerns of parents in North America, and no studies examining a process to improve pediatric lumbar puncture consent. Here the investigators conduct a randomized control study of a short educational video on a handheld device as an adjunct to the formal consent process.

Methods: 72 patients were enrolled, evenly divided between the control arm and video arm of the study. A survey was provided examining four key indices: parent self-rated understanding of the procedure, their perception of its safety, their perception of the painfulness and their overall comfort with their child undergoing LP. In addition, demographic characteristics such as prior experience with LP or epidural, language spoken at home, age of the child and indication for lumbar puncture, as well as qualitative information about parent concerns were collected.

ELIGIBILITY:
Inclusion Criteria:

* parent of a patient less than 17 years of age
* parent present for consent
* patient under the care of the neurology team (directly or consulting)
* consenting physician able to communicate with parent directly or through a translator

Exclusion Criteria:

* patients with emergent indications for lumbar puncture, such as bacterial meningitis
* parent's unable to communicate in English and no translator was available
* consent not performed in person (over the phone)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Likert Scale for Parent Understanding, Pain perception, Safety Perception and Comfort | within 10 minutes of consent discussion (controls) or viewing the video (video group)
  4 separate Likert scales from 1-10 (1 is low, 10 is high) for each of understanding of procedure, pain perception, safety perception and comfort with procedure, each individual scale will be reported. For understanding, safety and comfort, a higher score represents better outcome, for pain perception a lower score represents better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Singhal, MD MSc, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunbar M, Paton G, Singhal A. An Educational Video Improves Consent in Pediatric Lumbar Puncture: A Randomized Control Trial. Pediatr Neurol. 2019 Nov;100:74-79. doi: 10.1016/j.pediatrneurol.2019.04.014. Epub 2019 May 13. PMID 31201072